CLINICAL TRIAL: NCT06153004
Title: Improving Outcomes in Depression in Primary Care in a Low Resource Setting: Evidence From a Pilot Study
Brief Title: OptimizeD Pilot Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Harvard School of Public Health (HSPH) (Other); Massachusetts General Hospital (Other); Centre for Addiction and Mental Health (Other); Brigham and Women's Hospital (Other); Vanderbilt University (Other); All India Institute of Medical Sciences, Bhopal (Other); Sangath (Other)
Responsible Party: Principal Investigator, Vikram Patel, Paul Farmer Professor and Chair of the Department of Global Health and Social Medicine, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB20-2144-pilot; 1R01MH121632-01A1 (NIH)
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Depression; Depressive Disorder
MeSH Terms: conditions — Depression; Depressive Disorder | interventions — Antidepressive Agents

STUDY DESIGN:
Intervention Model Description: Fluoxetine versus a contextually adapted version of behavioral activation called the Healthy Activity Program (HAP) delivered by non-specialists for the treatment of depression
Who Masked: Outcomes Assessor
Masking Description: Masked (blinded) field-based assessors will conduct all outcome assessments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Activity Program (HAP) (Experimental): HAP is a brief psychological treatment adapted from behavioral activation therapy, an empirically supported psychological treatment recommended by the World Health Organization.
  Interventions: Behavioral: Healthy Activity Program (HAP)
- Antidepressant medication (ADM) (Experimental): Fluoxetine is a selective serotonin reuptake inhibitors (SSRIs) and one of the safest medications used to treat depression. It is a routinely used medication and part of the Essential Drug List (EDL) in India.
  Interventions: Drug: Antidepressant medication (ADM)

INTERVENTIONS:
Behavioral: Healthy Activity Program (HAP) — HAP, delivered over 6-8 sessions by non-specialist healthcare workers, has behavioural activation as the core psychological strategy along with other strategies such as problem-solving and activation of social networks.
  Arms: Healthy Activity Program (HAP)
Drug: Antidepressant medication (ADM) — Patients assigned to antidepressant medication will start on fluoxetine 20 mg/day which can be raised to 40 mg/day (the maximum mandated by treatment guidelines for primary care in India) at week 3 or 6 for patients who have yet to remit. Patients who cannot tolerate fluoxetine will be switched to escitalopram.
  Arms: Antidepressant medication (ADM)

SUMMARY:
This pilot study aims to explore and refine the trial procedures that will be implemented in a larger-scale clinical trial scheduled to commence in March 2024 (NCT05944926). As part of this study, 60 patients with moderate to severe depression will be randomized to either psychotherapy based on behavioral activation called the Healthy Activity Program (HAP) or antidepressant medication.

The pilot study has two primary objectives:

1. Evaluate the feasibility and acceptability of the study
2. Collect essential outcome data in preparation for the larger trial

DETAILED DESCRIPTION:
This pilot study will play a pivotal role in preparation for the forthcoming larger clinical trial, named the OptimizeD study, scheduled for launch in March 2024 (NCT05944926).

The primary objective of the OptimizeD study is to explore whether different patients respond differentially to a brief psychological treatment, known as the Healthy Activity Program, or a widely used generic Selective Serotonin Reuptake Inhibitor (fluoxetine). If such differences exist, this study aims to explore whether one can develop a machine learning-generated precision treatment rule to predict the most effective treatment based on individual baseline characteristics.

The pilot study has two primary objectives:

1. Evaluate the feasibility and acceptability of the study:

   This pilot study will focus on assessing the feasibility and acceptability of the research protocol, including recruitment strategies, data collection methods, interventions, and risk management procedures. This evaluation will help refine and tailor the study procedures and play a critical role in setting the stage for the subsequent OptimizeD study.
2. Collect essential outcome data in preparation for the larger trial:

This study will test and refine the data instruments, gather initial data on efficacy, and refine the baseline assessment (which will serve as the cornerstone for the development of the precision treatment rule).

ELIGIBILITY:
Inclusion Criteria:

* Participants will be adults aged 18 or over of any gender attending one of eight Primary Health Care Centers with a "diagnosis" of moderate to severe depression based on scores of 10 or above on the Patient Health Questionnaire-9 (PHQ-9).

Exclusion Criteria:

* Women who are pregnant or are breastfeeding or lactating
* Patients with a history of psychosis including schizophrenia spectrum disorders or bipolar disorder.
* Participants planning to move out of the study area during the follow-up period.
* Patients over 65 years of age with evidence of cognitive impairment - Patients who do not speak the study or local language (English or Hindi)
* Patients who are undergoing treatment for depression at the time of recruitment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by recruitment rate | 3-months
  The investigators will assess enrolment rate for eligible participants
Feasibility as measured by retention rate | 3-months
  The investigators will evaluate retention rates, which are calculated as the ratio of patients who complete the study to the total number of patients enrolled
Feasibility of study assessments | 3-months
  The investigators will examine adherence rates to study procedures and the barriers to study participation reported by participants over the course of the study.
Acceptability of interventions by participants | 3-months
  The investigators will assess treatment compliance. For the HAP arm, this will be defined as having completed at least six sessions. For the ADM arm, this will be defined as having completed more than 80% of the recommended 12-week course of antidepressant medication.

SECONDARY OUTCOMES:
Change from Baseline in Depressive Symptoms | 3-months
  The investigators will measure depressive symptoms using the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a 9-item self-report scale to screen for symptoms of depression. Items are rated on a 4-point Likert scale from 0 (not at all) to 3 (nearly every day), with total scores ranging from 0 to 27, where higher scores indicate more severe depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Sangath, Bhopal, Madhya Pradesh, India

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared through the National Institute of Mental Health (NIMH) Data Archive. To ensure participant privacy and data security, all shared data will be de-identified according to established protocols and guidelines. The data sharing plan will be periodically reviewed and updated, as necessary, to align with evolving best practices, policies, and guidelines for data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available indefinitely or for as long as the NIMH repositories support it.
Access Criteria: Researchers and interested parties who wish to access the data can submit a formal data access request to the NIMH Data Archive. Researchers who gain access to the data will be required to comply with the data usage policies and guidelines set forth by the NIMH Data Archive.
URL: https://nda.nih.gov/

REFERENCES:
- See also: Study description — https://mentalhealthforalllab.hms.harvard.edu/optimized